CLINICAL TRIAL: NCT05913375
Title: Stereotactic Management of Arrhythmia - Radiosurgery Treatment and Evaluation of Response in Ventricular Tachycardia
Acronym: SMARTER-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Leszek Giec Upper Silesian Medical Center of the Medical University of Silesia in Katowice, Poland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB/430-77/23
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-06

CONDITIONS: Ventricular Tachycardia
Keywords: radioablation; stereotactic arrhythmia radioablation (STAR); stereotactic body radiotherapy (SBRT); ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac radioablation (Experimental): Patients with ventricular tachycardia will undergo cardiac radiosurgery with one fraction of 20 Gy to the arrhythmia substrate, as determined by the electrophysiological cardiac mapping.
  Interventions: Radiation: Stereotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — Non-invasive delivery of ablative radiotherapy dose to the arrhythmia substrate defined with electroanatomical mapping (EAM)
  Other Names: Stereotactic Arrhythmia Radioablation, Cardiac Radiosurgery

SUMMARY:
Prospective single-arm study investigating the efficacy and safety of non-invasive cardiac radiosurgery for the treatment of ventricular tachycardia (VT) with reduced dose of radiation (20 Gy). The efficacy and safety outcome measures will be compared with historical control - patients treated within the SMART-VT study (NCT04642963) with a single dose of 25 Gy to test the hypothesis that reduced dose of radiation is similarly effective in terms of reduction of VT burden.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with structural heart disease
* Patients with implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy with defibrillation (CRT-D)
* Clinically symptomatic ventricular arrhythmia despite adequate treatment, with episodes of ventricular tachycardia occurring at least 3 times per month
* At least one episode of monomorphic ventricular tachycardia recorded during an electrophysiological examination
* Recurrent VT despite at least one previous failed attempt at percutaneous ablation or disqualification from this treatment method (eg, patients after percutaneous closure of patent foramen ovale, ventricular septal defect).
* Persistent recurrence of VT despite adequate pharmacotherapy.
* Informed consent of the patient to participate in the study.

Exclusion Criteria:

* Premature ventricular contractions
* Cardiac damage requiring inotropic treatment
* Implantation of left ventricular assist device (LVAD)
* Ventricular arrhythmia in the course of channelopathy
* Reversible cause of VT
* New York Heart Association (NYHA) stage IV heart failure
* Myocardial infarction or cardiac surgery in the last 3 months.
* Life expectancy less than 6 months
* Polymorphic ventricular tachycardia
* Pregnancy or breastfeeding
* Substrate location that prevents safe radiotherapy (eg due to location relative to critical organs, or dose given during previous radiotherapy treatments).
* Evidence of an active systemic, pulmonary or pericardial inflammatory process that has required systemic treatment in the past 6 months (eg disease-modifying drugs, steroids, immunosuppressants). Patients treated for sarcoidosis who are currently in remission on chronic immunosuppressive drugs, without current signs of an acute inflammatory process, may be included in the study.
* Active, uncontrolled malignancy and/or chemo/immunotherapy in the past month or planned within the month following radioablation.
* Lack of the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment | 6 months
  Number of patients with a reduction of the number of ventricular tachycardia (VT) episodes by at least 50% within 6 months after the irradiation compared to the number of VT episodes within 6 months before the intervention (based on registration from ICD/CRT-D), including:
  * the number of high-energy discharges
  * number of low-energy discharges for VT that was treated with stereotactic radiotherapy (STAR)

SECONDARY OUTCOMES:
Six-month survival without VT episodes | 6 months
Number of patients with complete elimination of ICD discharges | 12 months
Number of patients with a 90% reduction in the number of ICD discharges | 12 months
Number of hospitalizations due to VT episodes | 12 months
Recurrences outside the irradiated area | 12 months
  Number of patients who developed VT with a different morphology than specified during qualification for the procedure
Early treatment safety | 3 months
  Number of serious adverse events (SAE) in the first 3 months after the intervention
Long term treatment safety | 12 months
  Number of SAE episodes within 12 months after the intervention
Assessment of the intensity and dynamics of changes in biochemical parameters of myocardial damage. | 12 months
  Intensity and dynamics of changes in cardiac-related biochemical indices after treatment, like troponin, cardiac creatine kinase (MB-CK) concentration and
Evaluation of complications and mortality, including cardiac mortality and emergency hospitalizations during post-treatment follow-up | 12 months
Change in the need for antiarrhythmic drugs | 12 months
Evaluation of changes in the left ventricular ejection fraction | 12 months
Evaluation of changes in the morphology of the heart in the ultrasound examination | 12 months
Assessment of compliance of the results of additional imaging with the results of EAM | 3 months
  Correlation of data from electroanatomical mapping with the results of additional imaging studies (CT, echocardiogram, MRI if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Sławomir Blamek, MD, PhD, MBA, Principal Investigator — Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch; Wojciech Wojakwoski, MD, PhD, Principal Investigator — Professor Leszek Giec Upper Silesian Medical Center of the Medical University of Silesia in Katowice; Marcin Miszczyk, MD, PhD, Study Chair — Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch
Locations (2):
- Poland (2):
  - Maria Skłodowska-Curie National Research Institute of Oncology, Gliwice Branch, Gliwice
  - Professor Leszek Giec Upper Silesian Medical Center of the Medical University of Silesia, Katowice

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared within the European Standardized Treatment and Outcome Platform for Stereotactic Therapy Of Re-entrant tachycardia by a Multidisciplinary consortium (STOPSTORM). The intention to share the anonymized data with the consortium will be clearly explained, and a written consent will be obtained from each participant.
Supporting Information: Study Protocol, SAP, ICF